CLINICAL TRIAL: NCT00000433
Title: Anti-Tumor Necrosis Factor (TNFR:Fc) in Ankylosing Spondylitis
Brief Title: Blocking Tumor Necrosis Factor in Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: N01 AR92244; NIAMS-043
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2003-02

CONDITIONS: Spondylitis, Ankylosing
Keywords: Spondylitis; Etanercept; ENBREL; Tumor necrosis factor-alpha
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylitis

INTERVENTIONS:
Drug: Anti-Tumor Necrosis Factor

SUMMARY:
The Division of Rheumatology at University of California San Francisco is conducting a research study on the treatment of ankylosing spondylitis (AS) with a new therapy currently used for people with other forms of arthritis. The drug, called Enbrel (or etanercept), is a protein that is given twice weekly by injection underneath the skin. It blocks the action of tumor necrosis factor-alpha (TNF-alpha), a substance that may be involved in AS, rheumatoid arthritis, and other inflammatory conditions. We will randomly assign patients to receive either the drug or a placebo (inactive treatment) for 4 months. The results we will monitor include morning stiffness, spinal mobility, activities of daily life, and safety of the drug.

DETAILED DESCRIPTION:
In this Phase II clinical trial we will use tumor necrosis factor receptor p75 fusion protein (TNFR:Fc, or etanercept) to treat patients with ankylosing spondylitis (AS). TNFR:Fc is an antagonist of tumor necrosis factor (TNF), a cytokine that researchers have shown to play a possible role in disease pathogenesis of ankylosing spondylitis, rheumatoid arthritis, and vasculitis, as well as other inflammatory conditions.

TNFR:Fc consists of two molecules of the extracellular portion of the p75 receptor, each consisting of 235 amino acids. The two receptors are fused to the Fc portion of human IgG1, which consists of 232 amino acids. The gene fragments encoding the truncated TNFR and the Fc portion of human IgG1 are expressed in a Chinese hamster ovary cell line.

Recent observations from animal and human studies suggest that tumor necrosis factor-alpha (TNF-alpha) may play a role in disease activity in AS and other seronegative spondyloarthropathies. This study aims to test the efficacy of TNFR:Fc used in conjunction with standard medications in the treatment of AS. We will give patients either 25mg of TNFR:Fc or placebo subcutaneously twice a week for 4 months. Outcome measures will include measures of function, pain, morning stiffness, patient global assessment, and swollen joint count, as well as safety measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ankylosing spondylitis
* Acceptable stable treatments during study: oral glucocorticoids (less than or equal to 10 mg/d) and/or NSAIDs at recommended doses and/or one of the following options: methotrexate (less than or equal to 20.0 mg/week); sulfasalazine (less than or equal to 3 grams/d); azathioprine (less than or equal to 2 mg/kg/d); methotrexate and sulfasalazine combination at doses listed above; 6-mercaptopurine (less than or equal to 1.5 mg/kg/d)

Exclusion Criteria:

* Diagnosis of psoriatic arthritis, inflammatory bowel disease, reactive arthritis, or Behýet disease
* Significant medical problems, such as diabetes mellitus
* History of active or recurrent infections
* Complete ankylosis of the entire spine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 1999-10; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: John C. Davis, MD, MPH, Principal Investigator — Division of Rheumatology, University of California - San Francisco Department of Medicine
Locations (1):
- UCSF-Clinical Trials Center, San Francisco, California, United States

REFERENCES:
- [Background] Gorman JD, Sack KE, Davis JC Jr. Treatment of ankylosing spondylitis by inhibition of tumor necrosis factor alpha. N Engl J Med. 2002 May 2;346(18):1349-56. doi: 10.1056/NEJMoa012664. PMID 11986408
- [Background] Davis JC Jr, Van Der Heijde D, Braun J, Dougados M, Cush J, Clegg DO, Kivitz A, Fleischmann R, Inman R, Tsuji W; Enbrel Ankylosing Spondylitis Study Group. Recombinant human tumor necrosis factor receptor (etanercept) for treating ankylosing spondylitis: a randomized, controlled trial. Arthritis Rheum. 2003 Nov;48(11):3230-6. doi: 10.1002/art.11325. PMID 14613288
- [Background] Davis JC Jr, Huang F, Maksymowych W. New therapies for ankylosing spondylitis: etanercept, thalidomide, and pamidronate. Rheum Dis Clin North Am. 2003 Aug;29(3):481-94, viii. doi: 10.1016/s0889-857x(03)00028-0. PMID 12951863